CLINICAL TRIAL: NCT05838703
Title: Comparing the Acute Effects of Tiotropium Handihaler With Tiotropium Respimat on the Ventilation Distribution in COPD Patients
Brief Title: Tiotropium Handihaler vs. Tiotropium Respimat in COPD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely due to funding, prior to enrollment of first participant
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Yuh Chin T Huang, MD, MHS, Principal Investigator, Duke University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00112737
Record Dates: First submitted 2023-03-24; First posted 2023-05-01 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tiotropium bromide (Spiriva Respimat) (Experimental): Images obtained using 129XeMRI will be obtained after one-time use of Spiriva Respimat
  Interventions: Drug: tiotropium bromide (Spiriva Respimat); Drug: Hyperpolarized 129XeMRI
- Tiotropium bromide inhalation powder (Spiriva HandiHaler) (Active Comparator): Images obtained using 129XeMRI will be obtained after one-time use of Spiriva HandiHaler
  Interventions: Drug: tiotropium bromide inhalation powder (Spiriva HandiHaler); Drug: Hyperpolarized 129XeMRI

INTERVENTIONS:
Drug: tiotropium bromide inhalation powder (Spiriva HandiHaler) — Spiriva HandiHaler is a COPD medication that is available for use.
  Arms: Tiotropium bromide inhalation powder (Spiriva HandiHaler)
Drug: tiotropium bromide (Spiriva Respimat) — Spiriva Respimat is a COPD medication that is available for use.
  Arms: Tiotropium bromide (Spiriva Respimat)
Drug: Hyperpolarized 129XeMRI — Xe129 hyperpolarized with use of MRI for evaluation of lung ventilation has recently been FDA approved

SUMMARY:
The purpose of this study is to determine if tiotropium Respimat will result in better ventilation distribution of the lung in COPD participants quantified by hyperpolarized XeMRI. This study is designed to simulate the real-life clinical setting where patients receive one-time instruction on the inhaler use.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients of either gender, age > 40.
2. Willing and able to give informed consent and adhere to visit/protocol schedules. (Consent must be given before any study procedures are performed)
3. Women of childbearing potential must have a negative urine pregnancy test. This will be confirmed before participation in this investigational protocol.
4. Clinical diagnosis of COPD confirmed by post-bronchodilator spirometry demonstrating FEV1/FVC < 0.70 in all GOLD stages (http://www.goldcopd.org/).
5. Patients who are tiotropium naïve or whose tiotropium can be withheld for 2 weeks before screening visit/visit 1

   Exclusion Criteria:
6. Upper respiratory tract infection within 6 weeks (in this case, we will re-screen the patient after 6 weeks)
7. 24/7 oxygen use
8. Previous history of pneumothorax
9. Evidence of interstitial, occupational or chronic infectious lung disease by imaging studies
10. For women of child bearing potential, positive pregnancy test.
11. Major chronic illnesses which in the judgement of the study physician would interfere with participation in the study
12. History of claustrophobia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Assess the change in ventilation distribution parameters by 129Xe MRI in patient while taking Spiriva HandiHaler | 1 visit, up to 4 hours
  Perform Pre- and Post-Spirometry with Spiriva HandiHaler to assess the ventilation distribution percentage in patients (no ventilation/total ventilation) while taking Spiriva HandiHaler
Assess the change in ventilation distribution parameters by 129Xe MRI in patient while taking patient while taking Spiriva Respimat | 1 visit, up to 4 hours
  Perform Pre- and Post-Spirometry with Spiriva Respimat to assess the ventilation distribution percentage in patients (no ventilation/total ventilation) while taking Spiriva Respimat
Assess the changes in Pre- and Post-Spirometry procedure while on Spiriva HandiHaler | 1 visit, up to 4 hours
  Perform Pre- and Post-Spirometry to examine the changes in FEV1/FVC
Assess the changes in Pre- and Post-Spirometry procedure while on Spiriva HandiHaler | 1 visit, up to 4 hours
  Perform Pre- and Post-Spirometry to examine the changes in FEV1
Assess the changes in Pre- and Post-Spirometry procedure while on Spiriva HandiHaler | 1 visit, up to 4 hours
  Perform Pre- and Post-Spirometry to examine the changes in FVC
Assess the changes in Pre- and Post-Spirometry procedure while on Spiriva HandiHaler | 1 visit, up to 4 hours
  Perform Pre- and Post-Spirometry to examine the changes in FEF25-75
Assess the changes in Pre- and Post-Spirometry procedure while on Spiriva Respimat | 1 visit, up to 4 hours
  Perform Pre- and Post-Spirometry to examine the changes in FEV1/FVC
Assess the changes in Pre- and Post-Spirometry procedure while on Spiriva Respimat | 1 visit, up to 4 hours
  Perform Pre- and Post-Spirometry to examine the changes in FEV1
Assess the changes in Pre- and Post-Spirometry procedure while on Spiriva Respimat | 1 visit, up to 4 hours
  Perform Pre- and Post-Spirometry to examine the changes in FVC
Assess the changes in Pre- and Post-Spirometry procedure while on Spiriva Respimat | 1 visit, up to 4 hours
  Perform Pre- and Post-Spirometry to examine the changes in FEF25-75